CLINICAL TRIAL: NCT03225599
Title: Cranial Osteopathic Manipulative Medicine as an Adjunct Treatment for Concussion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwell Health (Other)
Collaborators: University of Pittsburgh Medical Center (Other)
Responsible Party: Principal Investigator, Rosanna C. Sabini, DO, Assistant Professor, Northwell Health
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Concussion COMM
Record Dates: First submitted 2017-07-14; First posted 2017-07-21 (Actual); Results first posted 2019-06-06 (Actual); Last update posted 2019-06-25 (Actual); Status verified 2019-06

CONDITIONS: Concussion Injury of Cerebrum; Cranial Osteopathic Medicine
MeSH Terms: conditions — Brain Concussion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Procedure (Experimental)
  Interventions: Other: Cranial Osteopathic Manipulative Medicine

INTERVENTIONS:
Other: Cranial Osteopathic Manipulative Medicine — The hands will be placed on the head using the "vault hold" (bilateral thumbs are off the head, index fingers on the temporal bones, middle fingers on the sphenoid bones, ring fingers on the mastoid and the 5th fingers on the occipital bone). Diagnosis and treatment of restrictions palpated on the scalp will be made using this hand position

SUMMARY:
Patients who have concussions exhibit an array of symptoms, also known as post-concussive symptoms, including headaches, feeling slowed down or foggy and difficulty with concentration. This study aims to determine if cranial osteopathy can provide additional or expedited symptom relief when accompanying current conventional treatments. The patients will be identified through routine clinical contact. If patients are found to be eligible and agree to participate, they receive a single session of cranial osteopathy in addition to their usual care through the concussion program.

ELIGIBILITY:
Inclusion Criteria:

* Concussion occurred within 8 weeks
* Age greater or equal to 14 years
* Complains of post-concussive symptoms with a symptom score of >10 on PCSS

Exclusion Criteria:

* Concussion occurred > 8 weeks
* Age less than 14 years
* Surgery of the cervical and/or thoracic spine within the last 3 months
* Currently receiving or has received workers compensation within the last 3 months
* Currently or potentially become involved in litigation related to the injury
* Received osteopathic craniosacral treatments within the last 3 months
* History of hydrocephalus, current infection or active tumor
* Active or marked depression, anxiety or psychosis

Min Age: 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2010-02-09 (Actual); Primary Completion 2010-06-30 (Actual); Study Completion 2013-01-26 (Actual)

RESULTS

PARTICIPANT FLOW:
Groups:
- Procedure: The treatment was performed with the patient lying comfortably in a supine position. The examiner's hand was initially placed at the occipito-atlantal junction of the top of the cervical spine to evaluate for fascial restrictions. Any palpated restrictions were released using a technique of myofascial release, where no passive or active range of motion was performed to the cervical region. Once the occipito-atlantal junction was determined to be free of restrictions, fingers were placed on the head using the Vault Hold (Figures 1 & 2). The Vault Hold was used for the administration of the procedure as is standard in osteopathic manipulative medicine by bilateral finger placement: thumbs are off the head, index fingers on the temporal bones, middle fingers on the sphenoid bones, ring fingers on the mastoid and the 5th fingers on the occipital bone. Each procedure lasted less than 30 minutes.
Period: Overall Study
Arm/Group | Procedure
Started | 9
Completed | 7
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | Procedure
Number analyzed (Participants) | 9
Age, Customized [Mean (Standard Deviation); unit: years] | 27.5 (16.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 4
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 9
Number of Participants that Underwent Procedure [Number; unit: participants] | 9

OUTCOME MEASURES:

1. Primary Outcome: Change in Concussive Symptoms on the Post Concussion Symptom Scale
Description: The Post Concussion Symptom Scale (PCSS) is a scale used to subjectively measure concussion symptoms. The minimum score is 0 and the maximum score is 132 (a maximum score of 6 for 22 items). The higher the value the worse the symptom. Twenty-two possible symptoms are graded and are the following:Headache, Nausea, Vomiting, Balance Problems, Dizziness, Lightheadedness, Fatigue, Trouble falling asleep, Sleeping more than usual, Sleeping less than usual, Drowsiness, Sensitivity to light, Sensitivity to noise, Irritability, Sadness, Nervous/Anxious, Feeling more emotional, Numbness or tingling, Feeling slowed down, Feeling like "in a fog," Difficulty concentrating, Difficulty remembering, and/or Visual problems. Total score can range from 0 to 132. Units of a scale is used.
Time Frame: 2 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Procedure
Number analyzed (Participants) | 9
units on a scale | 9 (7)

ADVERSE EVENTS:
Time Frame: 2months
Description: There were no direct adverse events.
Arm/Group | Procedure
All-Cause Mortality (participants affected / at risk) | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9
Other Adverse Events (participants affected / at risk) | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes